CLINICAL TRIAL: NCT00716157
Title: A Prospective Study to Evaluate the Incidence and Patterns of Nausea and Vomiting in Patients Receiving Combined Chemotherapy and Radiation
Brief Title: Incidence and Patterns of Nausea/Vomiting With Combined Chemotherapy and Radiation
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 04C.466; 2004-16 (Other: CCRRC); 1002004024 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Cancer of the Head and Neck; Cancer of the Lung; Cancer of the Esophagus; Gastro-esophageal Junction Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Adult patients receiving both radiation therapy and chemotherapy

SUMMARY:
Questionnaire study to observe the incidence and pattern or nausea and vomiting in patients receiving combined chemotherapy and radiation. 83% of patients experience radiation therapy-induced vomiting; significant nausea and vomiting could develop with concurrent chemotherapy despite standard anti-nauseous medication prophylaxis.

DETAILED DESCRIPTION:
Questionnaires will be answered daily on a weekly basis during period of radiation and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Concurrent radiation and chemotherapy treatment
* Aerodigestive malignancy

Exclusion Criteria:

* Other causes of vomiting (i.e.gastrointestinal obstruction...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University practice patients with aerodigestive malignancy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Assess incidence and patterns of nausea and vomiting in patients undergoing concurrent chemotherapy and radiation | week of treatment

SECONDARY OUTCOMES:
Assess the impact of nausea and vomiting on the patients' daily functioning | week of treatment
Study the incidence of mucositis and esophagitis | week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rita Axelrod, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States